CLINICAL TRIAL: NCT01128712
Title: An Open Label, Randomized Study Prospectively Examining the Effect on Anxiety in Partial Epilepsy Patients Treated With Pregabalin
Brief Title: Effect on Anxiety in Partial Epilepsy Patients Treated With Pregabalin
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of enrollment. terminated in 2014. no data analysis.
Sponsor: Northeast Regional Epilepsy Group (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Evan Fertig, Director of Research, Northeast Regional Epilepsy Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEREG-001
Record Dates: First submitted 2010-05-20; First posted 2010-05-24 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Epilepsy, Complex Partial
MeSH Terms: conditions — Epilepsy, Complex Partial | interventions — Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Other): Pregabalin (150mg/day)
  Interventions: Drug: Pregabalin
- Group 2 (Other): Pregabalin (450mg/day)
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Pregabalin — 150 mg /day
  Other Names: Lyrica
  Arms: Group 1
Drug: Pregabalin — 450 mg/day
  Other Names: Lyrica
  Arms: Group 2

SUMMARY:
To prospectively demonstrate the superior anxiolytic effect of high dose pregabalin (PGB) therapy (450 mg/day) compared to low dose PGB therapy (150 mg/day) in subjects with medically refractory partial epilepsy not fully controlled despite treatment with 1-2 concomitant antiepileptic drugs (AEDs).

DETAILED DESCRIPTION:
Background

Interictal anxiety symptoms are reported in two-thirds of patients with epilepsy and represent an underrecognized and undertreated aspect of the disorder. Interictal anxiety is postulated to stem from both fear of seizure recurrence ("seizure phobia") and dispersed locus of control.In addition, anxiety and the most common forms of partial onset epilepsy are viewed to arise from dysfunction in a common neurobiological substrate-the amygdala and other structures within the limbic system.

Background on Pregabalin

Pregabalin (CI-1008,Lyrica) is a chemical analogue of the mammalian neurotransmitter gamma-aminobutyric acid (GABA),although it does not bind to or activates GABA receptors or inhibit GABA uptake. Pregabalin is an alpha-2-delta ligand that has analgesic, anxiolytic, and antiepileptic activity.

Rationale

Antiepileptic drugs (AEDs) are commonly used for mood disorders including anxiety.Pregabalin (PGB) the most recently FDA-approved AED for add-on therapy for refractory partial seizures also has demonstrated efficacy in Generalized Anxiety Disorder. PGB binds to the alpha-2-delta subunit protein of voltage-gated calcium channels, and in animal models, has anxiolytic and anti-epileptic effects via pre-synaptic inhibition of the release of several excitatory neurotransmitters.

ELIGIBILITY:
Inclusion Criteria

* An IRB-approved consent form signed and dated by the subject
* A diagnosis of partial epilepsy which is drug resistant according to the International League Against Epilepsy criteria (Failure of adequate trials of two tolerated and appropriately chosen and used AED schedules (whether as monotherapies or in combination) to achieve sustained seizure freedom). Furthermore to meet the ILAE definition of drug resistance, subjects will have had breakthrough seizures occurring at a frequency of less than 3 times the longest pretreatment interseizure interval or every 12 months, which ever is longer.
* Subjects that score ≥18 on Beck Anxiety Inventory will be included in the study
* Subjects from 18 to 75 years, both inclusive.
* Females without childbearing potential or childbearing potential using medically accepted forms of birth control (pre-menarcheal, post-menopausal, bilateral oophorectomy or tubal ligation, complete hysterectomy, or medically accepted form of contraception).
* Subject judged by the Investigator to be reliable and capable of adhering to the protocol, visit schedules, and able to understand and complete study instruments.
* CT or MRI scan performed within 2 years of screening and without evidence of a progressive lesion or neurological condition.
* Electroencephalogram consistent with partial epilepsy and does not demonstrate generalized spike wave.
* Currently treated with a stable dose of 1-2 AEDs for a minimum of 4 weeks (3 months for phenobarbital and primidone). Benzodiazepines used as a rescue therapy for seizures and used no more than once a week will be permitted.

Exclusion Criteria

* History of psychogenic non-epileptic seizures.
* The subject is pregnant or lactating.
* Women with reproductive potential who refuse to use medically accepted forms of birth control.
* Presence of any clinically significant laboratory abnormality which in the judgement of the investigator should exclude the subject from the study.
* Presence of any progressive, demyelinating, or degenerative neurological condition.
* Subject is currently taking gabapentin.
* History of an allergic reaction to gabapentin or PGB.
* History of worsened seizures or serious adverse reactions to gabapentin.
* History of suicide attempt.
* No active suicidal plan/intent or active suicidal thoughts in the last 6 months.
* Current use or use within the previous three months prior to screening of antidepressant, anxiolytic, or antipsychotic agents. Subjects using benzodiazepines for anxiety will not be permitted.
* Diagnosis of Bipolar Disorder, Schizophrenia, psychotic disorder (excluding post-ictal psychosis), Major Depression requiring hospitalization in the past 2 years, or other psychological or behavioral condition which in the judgement of the investigator should exclude the subject from the study.
* A history of alcoholism, drug abuse, or drug addiction within the last 2 years.
* Any contraindication to use of PGB.
* Any clinical condition (e.g. severe renal impairment, chronic hepatic disease, serious infection, and or bone marrow depression) which will impair participation in the trial.
* History of multiple drug allergies or severe drug allergy.
* Subjects with vagal nerve stimulators (VNS).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change in Beck Anxiety Score | week 0 - week 6
  The primary outcome variable will be the change in the Beck Anxiety Inventory (BAI) score as measured at the baseline and final visits.

SECONDARY OUTCOMES:
Change in BDI , NHS3 , STAI , NDDI-E and seizure frequency | week 0 - week 6
  The secondary outcome variables will be the change in the Beck Depression Inventory, change in National Hospital Seizure Severity Scale (NHS3) score, change in seizure frequency, change in Stait-Trait Anxiety Scale (STAI),and change in the National Disorders Depression Inventory for Epilepsy Screening Tool (NDDI-E) as measured at the baseline and final visits.

CONTACTS AND LOCATIONS:
Overall Officials: Evan Fertig, MD, Principal Investigator — Northeast Regional Epilepsy Group
Locations (1):
- Northeast Regional Epilepsy Group, Hackensack, New Jersey, United States